CLINICAL TRIAL: NCT04195243
Title: Acute Effect of Dapagliflozin vs Empagliflozin Administration on Flow Mediated Dilation in Patients With Type 2 Diabetes Mellitus
Brief Title: Dapagliflozin vs Empagliflozin on Flow Mediated Dilation in Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Centro Universitario de Ciencias de la Salud, Mexico (Other)
Responsible Party: Principal Investigator, Fernando Grover Paez, Investigador Principal, Centro Universitario de Ciencias de la Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CUCS-INTEC-MV-HADES-001
Record Dates: First submitted 2019-12-04; First posted 2019-12-11 (Actual); Last update posted 2019-12-11 (Actual); Status verified 2019-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Dapagliflozin; Empagliflozin; FMD; T2DM; Endothelial disfunction
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin; empagliflozin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dapagliflozin (Experimental): Individuals with T2DM controlled with metformin; with no hypertension neither treated with insulin.
  Dapagliflozin capsules, 10 mg 1 time daily 5 minutes before the first meal
  Interventions: Drug: Dapagliflozin Pill
- Empagliflozin (Experimental): Individuals with T2DM controlled with metformin; with no hypertension neither treated with insulin.
  Empagliflozin capsules, 25 mg 1 time daily 5 minutes before the first meal
  Interventions: Drug: Empagliflozin Pill
- Placebo (Placebo Comparator): Individuals with T2DM controlled with metformin; with no hypertension neither treated with insulin.
  Dapagliflozin capsules, 400 mg 1 time daily 5 minutes before the first meal
  Interventions: Drug: Placebo pill

INTERVENTIONS:
Drug: Dapagliflozin Pill — The patient will take one pill, every 24 hr, during 7 days
  Other Names: Forxiga; Dapagliflozin
  Arms: Dapagliflozin
Drug: Empagliflozin Pill — The patient will take one pill, every 24 hr, during 7 days
  Other Names: Jardiance; Empagliflozin
  Arms: Empagliflozin
Drug: Placebo pill — The patient will take one pill, every 24 hr, during 7 days
  Other Names: Calcined magnesia
  Arms: Placebo

SUMMARY:
Type 2 diabetes mellitus (T2DM) is a considered one of the main global health challenges; the vascular endothelium plays an important role in vascular dysfunction in DM; Hyperglycemia induced by it is recognized as the main factor for the development of vascular complications of the disease, secondary to a reduction in nitric oxide production; "flow-mediated dilation" is the most commonly used technique for the evaluation of endothelial function, being the non-invasive method most widely used. It has been reported that with the use of SGLT2 inhibitors the development of cardiovascular complications in patients with T2DM is a decrease, as well the arterial stiffness, endothelial dysfunction and increasing on the shear stress and blood viscosity; and experimentally.

DETAILED DESCRIPTION:
The objective of this study, is to evaluate the acute effect of the administration of dapagliflozin in comparison with the administration of empagliflozin on endothelial disfunction in individuals with T2DM; we will conduct a double-blind, randomized, placebo-controlled, trial with 3 groups, each group of 24 male and female patients, between 40-65 years of age with T2DM, without hypertension, treated with insulins or thiazide diuretics. Randomization will determine who will receive the intervention during 7-days trial (Empagliflozin 25 mg 1 time daily 5 minutes or Dapagliflozin 10 mg before the first bite of each meal or approved placebo capsules), the patients will also continue with their usual treatment. The clinical findings and laboratory test and laboratory test include a metabolic profile and biosafety, baseline and at 7 days. Body weight, body fat, body mass index (BMI) and blood pressure will be determined during the initial and final visit, likewise, hemodynamics parameters of endothelial disfunction by flow mediate dilation with a high-resolution UNEX EF38G® ultrasound. Adverse events to treatment will be documented. Statistical analysis: Mann-Whitney U Test and Wilcoxon exact test. A p <0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T2DM
* HbA1c > 7 y < 10
* BMI 25 - 34.9 kg/m2
* Signature of consent under information

Exclusion Criteria:

* Hypertension
* Treated with insulin and / or loop diuretics and thiazides
* T1DM
* Hypotension
* With any autoimmune disease
* Liver disease
* Women who do not have a safe method of contraception
* Women who are taking oral contraceptives or under treatment with hormone replacement therapy
* Woman pregnant or breastfeeding
* Untreated thyroid disease
* Patients with a cardiovascular disease that contraindicates the use of this pharmacological class
* Glomerular filtration rate <60ml/min (Cockcroft-Gault)

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-12-02 (Estimated); Primary Completion 2020-06-29 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Flow Mediated Dilation | 7 days
  Change from baseline Flow mediated dilation at 7 days. Using a high-resolution UNEX EF38G ultrasound®, in a room at 22°C, with the patient lying supine, and the right arm extended

SECONDARY OUTCOMES:
Fasting plasma glucose | 7 days
  Before and after intervention, using the BioSystems® Glucose Oxidase / Peroxidase kit; in an automated clinical chemistry analysis equipment brand XL-100Erba
Total cholesterol | 7 days
  Before and after intervention, using the BioSystems® Glucose Oxidase / Peroxidase kit.
Triglycerides | 7 days
  Before and after intervention, using the BioSystems® Glycerol phosphate Oxidase / Peroxidase kit.
High-density lipoprotein cholesterol | 7 days
  Before and after intervention, using the BioSystems® Direct / Detergent HDL kit
Low-density lipoprotein cholesterol | 7 days
  Before and after intervention using the BioSystems® Cholesterol Oxidase / Peroxidase kit
Creatinine | 7 days
  Before and after intervention the BioSystems® kit Modified Jaffe's no deproteinization
Blood pressure | 7 days
  Before and after intervention using an OMRON calibrated electronic digital sphygmomanometer model HEM 907 XL will be used. The patient will remain seated in a chair resting his back on the backrest, with a minimum rest of 5 minutes, The average of 3 measurements such as BP will be taken

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Grover Paez, PhD, Study Director — Institute of Experimental and Clinical Therapeutics (INTEC), CUCS
Locations (1):
- Institute of Experimental and Clinical Therapeutics (INTEC), CUCS, University of Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No